CLINICAL TRIAL: NCT02449967
Title: HepaSphere Interventional Therapy Using Digital Subtraction Angiography（DSA） for Pancreatic Cancer: Clinical Trial
Brief Title: HepaSphere Interventional Therapy Using Digital Subtraction Angiography（DSA） for Pancreatic Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pancreatic Cancer HepaSphere
Record Dates: First submitted 2015-05-12; First posted 2015-05-21 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2015-08

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; HepaSphere
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HepaSphere (Experimental): pancreatic cancer patients received HepaSphere interventional therapy using the digital subtraction angiography（DSA）
  Interventions: Procedure: interventional therapy
- control (No Intervention): pancreatic cancer patients did not receive any interventional therapy

INTERVENTIONS:
Procedure: interventional therapy — pancreatic cancer patients received HepaSphere interventional therapy using the digital subtraction angiography（DSA）
  Arms: HepaSphere

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of HepaSphere interventional therapy using digital subtraction Angiography（DSA）for pancreatic cancer.

DETAILED DESCRIPTION:
By enrolling patients with pancreatic cancer adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of HepaSphere interventional therapy using digital subtraction Angiography（DSA）for pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-80
2. Karnofsky performance status >60
3. Diagnosis of pancreatic cancer based on histology or the current accepted radiological measures.
4. Classification tumor,nodes,metastasis-classification(TNM) stage: Ⅱ,Ⅲ,Ⅳ
5. Will receive interventional therapy
6. Life expectancy: Greater than 3 months
7. Patients' routine blood test, liver function and kidney function have no obvious abnormalities
8. Ability to understand the study protocol and a willingness to sign a written informed consent document

Exclusion Criteria:

1. Patients with other primary tumor except pancreatic cancer
2. History of coagulation disorders or anemia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2018-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse events | 1 year

SECONDARY OUTCOMES:
Percentage of lesions that show no sign of recurrence 12 months after interventional therapy | 1 year
Progress free disease (PFS) | 1 year
Overall survival (OS) | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi Liu, PhD, Study Chair — Fuda Cancer Hospital
Locations (1):
- Central laboratory in Fuda cancer hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Niu L, Chen J, Yao F, Zhou L, Zhang C, Wen W, Bi X, Hu Y, Piao X, Jiang F, Zeng J, Liu W, Li J, He L, Mu F, Zuo J, Xu K. Percutaneous cryoablation for stage IV lung cancer: a retrospective analysis. Cryobiology. 2013 Oct;67(2):151-5. doi: 10.1016/j.cryobiol.2013.06.005. Epub 2013 Jun 24. PMID 23806858
- See also: related information — http://www.ncbi.nlm.nih.gov/pubmed/25937772